CLINICAL TRIAL: NCT06234371
Title: Financial Incentives for Therapy Completion: A Randomized Controlled Trial With U.S. Veterans
Brief Title: Financial Incentives for Veteran Therapy Completion
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Cronin (Other)
Collaborators: University of Georgia (Other)
Responsible Party: Sponsor-Investigator, Christopher Cronin, Assistant Professor, University of Notre Dame
Organization: University of Notre Dame (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-05-6633
Record Dates: First submitted 2024-01-02; First posted 2024-01-31 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Motivation; Stress Disorder; Post Traumatic Stress Disorder; Depression; Depressive Disorder
Keywords: Veterans; Outpatients; Counseling
MeSH Terms: conditions — Stress Disorders, Traumatic; Stress Disorders, Post-Traumatic; Depression; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: After participants give consent, they are enrolled in the study. Randomization will be done via the Qualtrics platform. The treatment group will be offered a $500 gift card for completing 6, 12, and 18 counseling sessions; up to $1,500 in total. Because RRC's practice involves prescribing and scheduling counseling in 6-session blocks, the financial awards are revealed to veterans in the treatment group in stages. After intake, treatment group individuals are told that they will receive a $500 gift card for completing the first 6 sessions. If the counselor decides that another 6-session block should be prescribed, then at the completion of the 5th session (i) the next 6 sessions are scheduled and (ii) the counselor reveals that the participant can earn another $500 for completing the 12th session. The same process takes place during session 11. Other than informing individuals in the treatment group of the gift cards, counseling services will not change as a result of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The treatment group will be offered a $500 gift card for completing 6, 12, and 18 counseling sessions; up to $1,500 in total. Because RRC's typical practice involves prescribing and scheduling counseling in 6-session blocks, the financial awards are revealed to veterans in the treatment group in stages. After intake, treatment group individuals are told that they will receive a $500 gift card for completing the first 6 sessions; later sessions and awards are not mentioned. If the counselor decides that another 6-session block should be prescribed, then at the completion of the 5th session (i) the next 6 sessions are scheduled (i.e., sessions 7 through 12) and (ii) the counselor reveals that the participant can earn another $500 for completing the 12th session. The same process takes place during session 11. As part of RRC's typical practice, no veterans are offered more than 18 sessions.
  Interventions: Behavioral: Financial Incentive
- Control (No Intervention): The control group will have access to the normal counseling services provided by RRC staff. Those in the control group will receive "business as usual" services offered by the RRC, which includes the same counseling services and evaluation of how many sessions an individual is recommended to receive.

INTERVENTIONS:
Behavioral: Financial Incentive — The intervention is offering a $500 gift card as an incentive for completing 6 counseling sessions to eligible individuals randomized into the treatment group. Another $500 gift card will be given after completing 12 counseling sessions, and another $500 gift card will be given after completing 18 counseling sessions.
  Arms: Treatment

SUMMARY:
Recovery Resource Council (RRC) is one of the largest and most comprehensive non-profit mental and behavioral healthcare providers in North Texas. Accredited by the Joint Commission in Behavioral Health and licensed by the State of Texas as an Outpatient Treatment Center, RRC strives to promote wellness and recovery through a variety of services and programming. An important component of RRC programming is providing free counseling services to hundreds of U.S. veterans annually. While RRC observes great success for veterans who complete counseling, attendance can be a major obstacle.

Veterans who approach RRC for individual counseling services and consent to participate will be randomly assigned to the treatment or control group. The control group will receive counseling as usual. The treatment group will receive $500 gift card payments upon completing their 6th, 12th, and 18th counseling sessions, i.e., $1,500 in gift cards for completing all 18 sessions, the usual prescribed length of therapy. Our primary focus is to examine the impact of the financial incentives on therapy attendance and attrition. In addition, the investigators will estimate the impact on mental health using mental health inventories collected over the course of therapy sessions.

DETAILED DESCRIPTION:
Study enrollment will occur starting in September 2023 and will continue through 2026. Veterans who are referred to RRC are subject to an eligibility screening via phone, during which time they must ensure that they are 18 years of age or older, hold veteran status, are deemed not suicidal by RRC staff, and will participate in individual counseling. Eligible veterans are then assigned an intake session time, during which they show any requested documentation, complete the standard RRC intake form, complete an initial mental health assessment, and go through the informed consent process with RRC staff. Any participant who does not want to participate in the study will still receive all services as usual. After a participant gives consent, they are enrolled in the study and complete additional intake questions via the Qualtrics platform. Randomization will be done through the Qualtrics platform, so that results can be communicated to veterans immediately during their intake session. Randomization odds will be 50-50. The investigators plan to enroll 600 individuals, of which approximately 300 individuals will be offered financial incentives for therapy.

The experimental portion of these procedures is the random assignment of individuals to be offered or to not be offered financial incentives for therapy. The treatment group will be offered a $500 gift card for completing 6, 12, and 18 counseling sessions; up to $1,500 in total. Because RRC's typical practice involves prescribing and scheduling counseling in 6-session blocks, the financial awards are revealed to veterans in the treatment group in stages. After intake, treatment group individuals are told that they will receive a $500 gift card for completing the first 6 sessions; later sessions and awards are not mentioned. If the counselor decides that another 6-session block should be prescribed, then at the completion of the 5th session (i) the next 6 sessions are scheduled (i.e., sessions 7 through 12) and (ii) the counselor reveals that the participant can earn another $500 for completing the 12th session. The same process takes place during session 11. As part of RRC's typical practice, no veterans are offered more than 18 sessions. The counseling received by the control group is identical to that of the treatment group, as is the scheduling of additional sessions.

During the consent process, participants consent to be followed in administrative records. The investigators will track several outcomes of interest as they become available using several sources:

1. A start-of-session mental health survey administered via Qualtrics. This survey pre-dates our study and is part of RRC's usual process.
2. An end-of-session survey on expected benefits and expected costs of continuing counseling administered via Qualtrics. These questions were designed by the researchers.
3. Clinical mental health screenings performed by the licensed therapists after 6, 12, and 18 sessions. The practice of collecting this information pre-dates our study and is part of RRC's usual process.

At the point that 300 individuals are enrolled in the study sample, the investigators plan to estimate the treatment effect to determine the feasibility of adding a third study arm. If the treatment effect on either average number of sessions completed or the probability of completing six sessions is sufficiently large and there is support from RRC to do so, the investigators plan to begin randomizing into a second treatment arm which will receive a gift card of value less than $500. If this third study arm becomes a reality, power calculations will be re-evaluated to shift to an updated optimal sample size.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participation requirements outlined in the informed consent form
* 18 years of age or older
* Holds veteran status
* Possesses and is willing to share SSN
* Possesses and is willing to share an active email address
* Individual is not screened out by RRC - i.e., RRC would agree to provide services independent of the research study
* Is participating in individual counseling

Exclusion Criteria:

* Individuals who are not interested in participating
* Individuals who do not consent
* Individuals posing a significant suicide risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2027-01-02 (Estimated); Study Completion 2028-01-02 (Estimated)

PRIMARY OUTCOMES:
Number of counseling sessions attended | 1 year following randomization
  Total number of counseling sessions attended
Completion of therapy | 1 year following randomization
  An indicator variable for completion of therapy will be constructed using discharge codes that RRC assigns to each patient. In particular, there is a discharge code for program completion (regardless of the number of sessions).

SECONDARY OUTCOMES:
Completion of every possible number of counseling sessions | 1 year following randomization
  e.g., at least 1 session, at least 2 sessions, etc. In other words, we will plot survival curves by treatment status.
Start-of-Session Mental Health Index and sub-components | 1 year following randomization
  Using the responses to start-of-session questions, investigators will create a summary standardized index of mental health at the start of each session.
Expected cost and benefit of therapy | 1 year following randomization
  Using the responses to survey questions asked at the end of each session regarding how a respondent thinks their symptoms will change after the next two sessions as well as how upsetting a respondent expects the next two sessions will be, investigators will create indicator variables corresponding to the categories of these expectations.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cronin, PhD, Principal Investigator — University of Notre Dame; Ethan Lieber, PhD, Principal Investigator — University of Notre Dame; Meghan Skira, PhD, Principal Investigator — University of Georgia
Locations (3):
- United States (3):
  - Recovery Resource Council East Campus, Dallas, Texas
  - Recovery Resource Council North Campus, Denton, Texas
  - Recovery Resource Council West Campus, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT06234371/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT06234371/ICF_001.pdf